CLINICAL TRIAL: NCT04913168
Title: Organizational Approaches to TWH for Low-Income Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Glorian Sorensen, Professor of Social and Behavioral Sciences, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TWH for Low Income Workers
Record Dates: First submitted 2021-05-25; First posted 2021-06-04 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Work-related Injury
Keywords: worker health; occupational safety and health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Experimental): Control Group; no intervention
  Interventions: Other: Front Line Worker Pilot Project
- Intervention Group (Experimental): Intervention Group; receives 13 month intervention
  Interventions: Other: Front Line Worker Pilot Project

INTERVENTIONS:
Other: Front Line Worker Pilot Project — 13-month intervention targeting workplace policies and programs focused on changes to safety and ergonomics, job enrichment, and work intensity for front line food service workers practices,

SUMMARY:
There is an urgent need for evidence-based interventions to reduce risk of musculoskeletal disorders (MSDs) and improve health and safety behaviors for low-income workers. Upstream interventions addressing these organizational characteristics and work experiences may be especially effective in preventing adverse health outcomes because they address underlying sources of elevated risk particularly important for low-wage workers. Low-wage workers have less schedule control, more irregular working hours, and shortened breaks due to time pressure to complete work tasks. The objective is to develop and test feasible intervention methods to modify the work organization and contribute to reductions in MSD risk, and improvements work-related well-being and job satisfaction. First, this study will identify characteristics of the work organization that can be feasibly modified through changes in management practices, based on interviews with food service managers and focus groups with workers. Second, the investigators will determine the feasibility and potential efficacy of an integrated TWH intervention in improving workers' ergonomic practices, MSD symptom, as well as in changing the work organization and environment related to work-related well-being and job satisfaction.

The contribution of this study will be significant because it is expected to contribute to reducing disparities in these health outcomes by directly intervening on an underlying source of these disparities.

DETAILED DESCRIPTION:
The food service industry employs 9.5 million workers in the U.S, many of whom are at elevated risk for a range of poor health outcomes. NIOSH's Total Worker Health™ (TWH) Program provides an innovative approach for addressing the shared pathways in the work organization and environment that impact both MSD risk and health and safety behaviors. This study takes advantage of an unusual opportunity to demonstrate the impact of changes in the work organization in collaboration with an industry partner that has committed to making such changes in concert with this study. Our central hypothesis is that an intervention targeting the work organization, as well as the work environment will show promising improvements in MSD outcomes and improvements in work-related well-being and job satisfaction.

The Specific Aims of this study include:

1. Identify factors in the work organization, expected to be associated with MSD risk and work-related well-being and job satisfaction, which can be feasibly modified through changes in management practices. The investigators will conduct formative research using qualitative data from workers and managers to explore two overarching issues to inform intervention development specific to this setting: (a) What work organizational factors do workers perceive as priorities for their safety and health? (b) What factors in the work organization do worksite and district managers believe can be feasibly modified through changes in policies and practices? The investigators will additionally explore barriers and facilitators to these changes, and factors contributing to sustainability.
2. Determine the feasibility and potential efficacy of an integrated TWH intervention designed to improve the work organization and environment, workers' MSD symptoms, ergonomic practices, and work-related well-being and job satisfaction. To provide the next level of evidence and prepare for a full-scale randomized control trial (RCT), the investigators will conduct a proof-of-concept (PoC) trial to evaluate an integrated TWH intervention in ten food service worksites randomly assigned to intervention and control conditions, to: (a) assess the feasibility of intervention delivery and the acceptability of the intervention; and (b) provide preliminary estimates of baseline levels, change from baseline to final, and intra-class correlation. The investigators will explore the working hypothesis that between pre- and post-intervention, compared to workers in control worksites, workers in intervention sites will report greater improvements in the primary outcomes, including ergonomic practices and MSD symptoms, work-related well-being and job satisfaction; and secondary outcomes, including improvements in the work organization and environment.

This PoC intervention will be tested in10 food service worksites randomly assigned to intervention and control. The 13-month intervention will target changes in the organizational and physical work environment and management practices, and supporting safe ergonomic practices and factors related to work-related wellbeing and job satisfaction. The investigators will compare differences between intervention and control sites in changes between pre- and post-intervention in worker health and safety behaviors and MSD symptoms through surveys of workers, and in the work organization and environment through manager surveys and on-site walk-through's. A rigorous process evaluation will be used to assess intervention feasibility. The contribution of this study will be significant because it is expected to contribute to reducing disparities in these health outcomes by directly intervening on an underlying source of these disparities.

ELIGIBILITY:
Inclusion Criteria:

* All front line workers including chefs, cooks, food preparers, servers, dishwashers, and cashiers

Exclusion Criteria:

* Front Line workers with supervisory responsibilities

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Change in Reduction in Pain and Injuries Worker Survey | 13 months
  Nordic Scale
Change in Improvements in Front Line Worker Turnover Intention Worker Survey | 13 months
  Turnover Intention Scale
Change in Improvement in Front Line Worker Well Being Worker Survey | 13 months
  WHO Wellbeing Scale

CONTACTS AND LOCATIONS:
Overall Officials: Glorian Sorensen, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sorensen G, Peters SE, Nielsen K, Stelson E, Wallace LM, Burke L, Nagler EM, Roodbari H, Karapanos M, Wagner GR. Implementation of an organizational intervention to improve low-wage food service workers' safety, health and wellbeing: findings from the Workplace Organizational Health Study. BMC Public Health. 2021 Oct 16;21(1):1869. doi: 10.1186/s12889-021-11937-9. PMID 34656090